CLINICAL TRIAL: NCT06710756
Title: A Phase I/IIa Image-Guided, Alpha-Particle Therapy Study of [203Pb]Pb-PSV359 and [212Pb]Pb-PSV359 in Patients With Solid Tumors That Are Known to be Fibroblast Activation Protein (FAP)-Positive
Brief Title: Lead-212 PSV359 Therapy for Patients With Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Perspective Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PSV359-001
Record Dates: First submitted 2024-11-25; First posted 2024-11-29 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Gastric Cancer; Esophageal Cancer; Colorectal Cancer; Ovarian Cancer; Head and Neck Cancer; Sarcoma; Mesothelioma
Keywords: Fibroblast Activation Protein; Solid tumor malignancy; Gastric cancer; Esophageal cancer; Colorectal cancer; Ovarian cancer; Head and neck cancer; Theronostic; Radiopharmaceutical; Radiotherapy; Alpha Particle; Pb-203; Pb-212
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms; Colorectal Neoplasms; Ovarian Neoplasms; Head and Neck Neoplasms; Sarcoma; Mesothelioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental): * Enrolled subjects are administered [203Pb]Pb-PSV359 (7mCi) for imaging FAP-expressing cancers.
  * Approximately Four cohorts of [212Pb]Pb-PSV359 dose levels will be explored for determining Recommended Phase 2 Dose (RP2D). Study subjects will be assigned to cohorts sequentially.
  Interventions: Drug: [203Pb]Pb-PSV359; Drug: [212Pb]Pb-PSV359
- Dose Expansion (Experimental): * Enrolled subjects are administered [203Pb]Pb-PSV359 (7mCi) for imaging FAP-expressing cancers.
  * Enrolled subjects are administered [212Pb]Pb-PSV359 (RP2D determined previously) for treatment of FAP-expressing cancers
  Interventions: Drug: [203Pb]Pb-PSV359; Drug: [212Pb]Pb-PSV359

INTERVENTIONS:
Drug: [203Pb]Pb-PSV359 — [203Pb]Pb-PSV359 is administered by intravenous bolus injection for single-photon emission computed tomography imaging.
Drug: [212Pb]Pb-PSV359 — [212Pb]Pb-PSV359 is administered by intravenous infusion for treatment of FAP expressing cancers.

SUMMARY:
Phase I/IIa image-guided, alpha-particle therapy study of [203Pb]Pb-PSV359 and [212Pb]Pb-PSV359 in patients with solid tumors that are known to be Fibroblast Activation Protein (FAP)-positive.

DETAILED DESCRIPTION:
This is a prospective, multi-center open label dose finding, dose expansion study of [212Pb]Pb-PSV359 in subjects with a positive Fibroblast Activation Protein (FAP) imaging scan with imaging agent.

FAP is specifically expressed on the surface of cancer-associated fibroblasts in some tumor tissues and therefore is an attractive target in the diagnosis and treatment of various cancers. Lead-212 ([212Pb]Pb-) based peptide-radiopharmaceuticals are an emerging class of targeted alpha-particle cancer therapies that have potential to improve delivery of a highly effective form of radiation.

This study will be conducted in 2 parts:

Part 1: Dose-escalation: [212Pb]Pb-PSV359 is administered in escalating doses to determine the Maximum Tolerated radioactivity (MTD) Dose and potential recommended Phase 2 dose (RP2D).

Part 2: Dose-expansion: This part will enroll subjects in expansion cohorts based on the identified MTD and RP2D for the selection of [212Pb]Pb-PSV359 doses for further clinical development.

A Dosimetry sub-set utilizing an imaging surrogate, [203Pb]Pb-PSV359, has been incorporated into the study in order to assess organ biodistribution and tumor uptake of the investigational products. This sub study will also estimate radiation dosimetry and correlate uptake of the investigation products with observed toxicities and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years
* Satisfactory organ function as determined by laboratory testing
* Eastern Cooperative Oncology Group performance (ECOG) status of 0 to 1
* Life expectancy > 3 months
* Progressive disease despite standard therapy or for whom no standard therapy exists
* Positive [203Pb]Pb-PSV359 SPECT/CT scan showing uptake of [203Pb]Pb-PSV359 in at least 1 known lesion on the 1-hour SPECT/ CT scan
* Histological, pathological, and/or cytological confirmation of solid tumor malignancy that is locally advanced or metastatic

Exclusion Criteria:

* Known hypersensitivity to the active agent or any of the excipients
* Active secondary malignancy
* Pregnancy or breastfeeding a child
* Known brain metastases
* Known active or uncontrolled infections requiring ongoing antifungals or antibiotics in the 3 days prior to enrollment
* Known medical condition which would make this protocol unreasonably hazardous for the patient
* Existence of any medical or social issues likely to interfere with study conductor that may cause increased risk to the subject or to others, e.g., lack of ability to follow radiation safety precautions
* Medical history of a condition resulting in a severe allergic reaction such as anaphylaxis or angioedema to known components of the investigational product or excipients
* Major surgery within 21 days prior to the administration of [212Pb]Pb-PSV359; the subject must be sufficiently recovered and stable before treatment administration
* Diagnosis of deep vein thrombosis or pulmonary embolism within 4 weeks prior to enrollment into the study
* Current abuse of alcohol or illicit drugs
* Treatment with any live/attenuated vaccine in the 7 days prior to enrollment
* Previous treatment with any systemic anticancer therapy within 4 weeks prior to treatment on study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2032-05-28 (Estimated)

PRIMARY OUTCOMES:
Determination of safety and tolerability of [203Pb]Pb-PSV359 | 30 days (±1day) post dose
  Incidence and severity of treatment-related adverse events following a single administration of [203Pb]Pb-PSV359 is determined
Determination of safety and tolerability of [212Pb]Pb-PSV359 | Up to 3 years
  Incidence and severity of treatment-related adverse events following a single and each repeated administration of [212Pb]Pb-PSV359 is determined
To determine the recommended phase 2 dose of [212Pb]Pb-PSV359 | Up to approximately 6 months
  The recommended phase 2 dose as determined by cohort observations and review by the Safety Monitoring Committee

SECONDARY OUTCOMES:
Determination of duration of response following treatment with [212Pb]Pb-PSV359 | Up to 3 years
  Median duration of response for subjects receiving at least 1 administration of [212Pb]Pb-PSV359 is assessed by RECIST V1.1 criteria
Determination of progression free survival following treatment with [212Pb]Pb-PSV359 | Up to 3 years
  Progression free survival for subjects receiving at least 1 administration of [212Pb]Pb-PSV359 is assessed by RECIST V1.1 criteria
Determination of pharmacokinetic properties of [203Pb]Pb-PSV359 and [212Pb]Pb-PSV359 | Up to approximately 3 yrs
  Blood radioactivity pharmacokinetic parameter such as area under the plasma concentration versus time curve (AUC) is determined.
Determination of pharmacokinetic properties of [203Pb]Pb-PSV359 and [212Pb]Pb-PSV359 | up to approximately 3 years
  Blood radioactivity pharmacokinetic parameter such as peak plasm concentration (Cmax) is determined
Determination of pharmacokinetic properties of [203Pb]Pb-PSV359 and [212Pb]Pb-PSV359 | up to approximately 3 years
  Blood radioactivity pharmacokinetic parameter such as the time (Tmax) to reach the maximum concentration (Cmax) is determined
Estimation of biodistribution of 203Pb PSV 359 using SPECT/CT scans | Up to approximately 3 years
  Activity in tumor(s) and organs as percentage of injected dose is assessed

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Saint Louis University, St Louis, Missouri
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania